CLINICAL TRIAL: NCT05600062
Title: Assessment of the Effect of Neutral Endopeptidase Inhibition on Vascular Leak and Leukocyte Accumulation in a Human Cantharidin Blister Model
Brief Title: Influence of NEP Inhibition on Vascular Leak and Inflammation (NEPi-INFLAMMATION)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Collaborators: Medical Research Council (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 288749
Record Dates: First submitted 2022-10-03; First posted 2022-10-31 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: ARDS; endothelium; CNP; Acute lung injury
MeSH Terms: conditions — Respiratory Distress Syndrome; Acute Lung Injury

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo tablet to be taken three times a day for three days
  Interventions: Drug: Placebo
- Racecadotril (Experimental): Racecadotril 100 milligrams (mg) three times a day for three days
  Interventions: Drug: Racecadotril 100 milligram (MG) Oral Capsule

INTERVENTIONS:
Drug: Racecadotril 100 milligram (MG) Oral Capsule — Licensed NEP inhibitor
  Other Names: Tiorfan
  Arms: Racecadotril
Drug: Placebo — Placebo capsule
  Arms: Placebo

SUMMARY:
Acute Respiratory Distress Syndrome (ARDS) is a severe type of lung injury that affects 10% of patients admitted to Intensive Care Units worldwide, with an unacceptably high mortality of up to 48% in those with the most severe form of the condition. It is a complex and poorly understood syndrome that results in progressive failure of the lungs. Crucially, the inflamed lungs allow fluid to leak from the circulation into the airspace, so that patients' lungs fill with fluid - "drowning from the inside". As this condition progresses, the patient typically requires increasing amounts of oxygen and eventually, support from a ventilator. To date, there are no effective treatments for ARDS that can limit, stop or repair this process.

This research study is aiming to look at a naturally occurring substance produced by blood vessels, C-type natriuretic peptide (CNP). The investigators have evidence suggesting that CNP plays a role in maintaining the barrier provided by blood vessels that stops fluid leaking out into tissues. This is based on various studies done on CNP by the investigators research group that have established its widespread role in maintaining cells that line blood vessels and play a vital role in lungs' barrier function: the endothelium.

CNP is broken down in part by an enzyme called Neutral endopeptidase and therefore, drugs that inhibit this enzyme would result in increased CNP concentration and activity. If CNP does in fact strengthen the lungs' endothelial barrier, then this class of drug may benefit patients with ARDS. The aim of this experimental medicine study is to assess the effect of using the licensed NEP inhibitor Racecadotril, in a well-established, safe model of inflammation-induced skin blisters in healthy human volunteers to determine primarily whether the fluid accumulation i.e. leak, in these blisters is reduced by treatment with this drug.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female volunteers
2. BMI of 18-40 kg/m2
3. Aged 18-45
4. Volunteers who are willing to sign the consent form

Exclusion Criteria:

1. Healthy subjects unwilling to consent
2. Smokers
3. Known sensitivity to Racecadotril
4. History of any serious illnesses, including recent infections or trauma
5. A personal history of keloid scarring, or a family history of keloid scarring in a first degree relative with similar skin pigmentation
6. Subjects taking systemic medication (other than the oral contraceptive pill)
7. Subjects who are pregnant or any possibility that a subject may be pregnant, unless in the latter case a pregnancy test is performed with a negative result
8. Women who are breastfeeding
9. Subjects with recent or current antibiotic use
10. Subjects with a history of skins conditions.
11. Subjects with a history of allergic reaction to any topical application or history of angioedema
12. Subjects with any history of a blood-borne infectious disease such Hepatitis B or C virus, or HIV.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Equal number of males and females
Enrollment: 48 (Estimated)
Dates: Start 2023-08-24 (Actual); Primary Completion 2026-01-17 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Powered unpaired inter-patient comparison of change in blister fluid volume following Racecadotril or placebo administration. | 24 hours after application of cantharidin
Powered paired intra-patient comparison of change in blister fluid volume following Racecadotril or placebo admininstration. | 24 hours after application of cantharidin

SECONDARY OUTCOMES:
Powered comparison of sex differences in change in blister volume following Racecadotril or placebo administration. | End of study
Difference in concentration of blister fluid cytokines; specifically Interleukin (IL) -1β, IL-6, IL-8, IL-10, CXCL1, CXCL2, CCL5 and CCL2 in volunteers receiving Racecadotril compared to placebo. | 24 hours after application of cantharidin
Comparison of change in blister fluid leukocyte count following Racecadotril or placebo administration | 24 hours after application of cantharidin
Comparison of change in pro and anti-inflammatory mediators from blister fluid following Racecadotril or placebo administration | 24 hours after application of cantharidin
Comparison of change in plasma cGMP following oral Racecadotril or placebo administration | 24 hours after application of cantharidin

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Hobbs, Principal Investigator — Queen Mary University London
Locations (1):
- William Harvey Research Institute- Heart Centre, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Fully anonymised data will be shared with fellow researchers via conference presentation and via publication of the results in scientific journals. Data will be shared between the research team directly undertaking the research
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 6 months after publication
Access Criteria: Access requests can be made to the investigators by email